CLINICAL TRIAL: NCT02271776
Title: The Effects of Galactooligosaccharide (GOS) on Peripheral Insulin Sensitivity and Body Weight Control in Obese Adults With Impaired Glucose Homeostasis
Brief Title: GOS and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: METC 143026
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2015-10

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Insulin Sensitivity
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — 4'-galactooligosaccharide; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galactooligosaccharide (Active Comparator): 5g 3x per day for 12 weeks
  Interventions: Dietary Supplement: Galactooligosaccharide
- maltodextrin (Placebo Comparator): 3x per day for 12 weeks (isocaloric to intervention)
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: Galactooligosaccharide — The dietary fiber GOS will be supplemented in powder form to regular daily food intake three times per day for 12 weeks
  Arms: Galactooligosaccharide
Dietary Supplement: maltodextrin
  Arms: maltodextrin

SUMMARY:
Based on our hypothesis that orally administered GOS will be fermented into a SCFA pattern high in acetate and that this will lead to beneficial effects on human substrate and energy metabolism, we aim to address the following primary objective:

To investigate the effects of a 12-week supplementation of GOS on peripheral insulin sensitivity and body weight control in obese adults with impaired glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

Overweight/obese (BMI ≥ 28 kg/m2 < 40 kg/m2) insulin impaired men and post-menopausal women with impaired glucose tolerance (IGT: 2h plasma glucose during 75g OGTT 7.8-11.1 mmol/l) and/or impaired fasting glucose (plasma glucose ≥ 5.6 mmol/l) aged 45-70 years will be included in the study.

In addition, subjects have to be weight-stable for at least 3 months prior to participation (no change in bodyweight, i.e. < 3kg).

Exclusion Criteria:

* diabetes mellitus
* gastroenterological diseases or major abdominal surgery (allowed i.e.: appendectomy, cholecystectomy)
* lactose intolerance and other digestive disorders
* cardiovascular disease, cancer, liver or kidney malfunction (determined based on ALAT and creatinine levels, respectively)
* disease with a life expectancy shorter than 5 years
* abuse of products (alcohol consumption > 15 units/week, or any drugs)
* excessive nicotine use defined as >20 cigarettes per day

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
systemic insulin sensitivity | change from baseline at 12 week supplementation

SECONDARY OUTCOMES:
substrate oxidation and energy expenditure | change from baseline at 12 week supplementation
plasma markers of substrate and energy metabolism | change from baseline at week 1 and at 12 week supplementation
fecal and plasma SCFA concentrations | change from baseline at week 1 and at 12 week supplementation
fecal microbiota composition | change from baseline at week 1 and at 12 week supplementation
skeletal muscle and adipose tissue gen and protein expression | change from baseline at week 1 and at 12 week supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Department of Human Biology, Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Canfora EE, van der Beek CM, Hermes GDA, Goossens GH, Jocken JWE, Holst JJ, van Eijk HM, Venema K, Smidt H, Zoetendal EG, Dejong CHC, Lenaerts K, Blaak EE. Supplementation of Diet With Galacto-oligosaccharides Increases Bifidobacteria, but Not Insulin Sensitivity, in Obese Prediabetic Individuals. Gastroenterology. 2017 Jul;153(1):87-97.e3. doi: 10.1053/j.gastro.2017.03.051. Epub 2017 Apr 8. PMID 28396144